CLINICAL TRIAL: NCT01155505
Title: Phase Ib of CC-5013 and Paclitaxel in Patients With Advanced Solid Tumors
Brief Title: Lenalidomide and Paclitaxel in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southern Europe New Drug Organization (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S095LEPT01
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CC-5013 in combination with Paclitaxel (Experimental): Cohorts of 3 evaluable patients will initially be entered within each dose level, sequentially. In each dose level the second and third patient will enter 2 weeks after the first one. The second and third patient may be treated simultaneously, except if a DLT is reported in the first patient, in which case the second and third patient should be treated sequentially, at least one week apart.
  Dose escalation will be done when all the patients included in each DL will finish the first treatment cycle. Three additional patients will be sequentially entered (separated by one week each other) if one DLT is observed in cycle 1 among the first 3 patients entered within a dose level. If a DLT is observed in a second patient at this dose level, no further dose escalation will be allowed and the dose level will be considered the MTD.
  Once the RD (one level below the MTD) has been defined, additional patients (up to 12) will be treated in order to confirm the safety profile of the combination.
  Interventions: Drug: Lenalidomide (CC-5013)

INTERVENTIONS:
Drug: Lenalidomide (CC-5013) — CC-5013 given PO daily on D1-D14 every 21 days and Paclitaxel administered IV over 1 hour on d1 and 8 every 21 days until tumor progression or unacceptable toxicity

SUMMARY:
This is a dose finding, open-label, uncontrolled, dose-escalation trial to determine the maximum Tolerated Dose (MTD) of the combination of CC-5013 (Lenalidomide)and paclitaxel in patients with advanced solid tumors.

Other purposes of the study are:

1. Define the safety profile of the CC-5013 and paclitaxel given in combination
2. Define the pharmacokinetics of CC-5013 and paclitaxel given in combination
3. Define the pharmacodynamic effects of the combination by monitoring potential biomarkers of the different biological activities of each component of the regimen
4. Define the optimal biological dose (OBD) and the dose recommended (RD) for phase II studies in selected tumor types (breast, ovary, prostate, NSCLC)
5. Collect evidence of antitumor activity in selected tumor types

DETAILED DESCRIPTION:
The new immunomodulatory drugs (IMiD) derivatives of thalidomide (CC-5013 lenalidomide and CC4047 pomalidomide) are endowed of direct antitumor activity besides the indirect effects attributed to antiangiogenic, antiinflammatory and T-cell co-stimulatory properties.

Combination therapy with cytotoxic agents or other anticancer drugs could lead to additive or synergistic interactions and support their clinical development in tumor types in which the specific activities of IMiDs could be of potential value.

Combinations with weekly paclitaxel could be of interest because of its antiangiogenic activity, antitumor activity in prostate, NSCLC, ovary, breast cancer, tumor types in which IMiD could be of clinical value because of either enhancement of tumor specific immunity (ovary, prostate) or inhibition of Treg function (breast, NSCLC, ovary).

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological diagnosis of solid tumors for which a treatment with paclitaxel could be indicated (preferentially ovary, breast, prostate, NSCLC)
* Documented progression of the tumor in the 3 months preceding the study
* Expected survival ≥ 3 months
* Age 18-75 years
* ECOG PS 0-1
* measurable/evaluable disease during escalation phase, according to modified RECIST criteria. For patients with ovarian and prostatic cancer, tumor markers (CA125 for ovarian and PSA for prostatic) are accepted as only evidence. Measurable/evaluable disease is mandatory during the RD expansion phase

  •≤ 2 prior lines of chemotherapy for metastatic disease. For ovarian patients reintroduction of a platinum at relapse, after an initial response lasting > 6 months is considered one chemotherapy regimen only
* Adequate contraception for all fertile patients
* Adequate hematological function as defined by: ANC ≥ 1.5 x 109/L, platelet count ≥100 x 109/L, hemoglobin ≥ 10 g/dL.
* Normal PTand INR; fibrinogen > lower Normal Limit (LNL)
* Adequate renal function, as defined by: creatinine ≤ 1.5 x UNL
* Adequate hepatobiliary function, as defined by the following baseline liver function tests:

  * total serum bilirubin within upper normal limit (UNL)
  * alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤2.5xUNL or ≤ 5xUNL in case of liver metastases; alkaline phosphatase (AP) ≤ 2.5xUNL. If total alkaline phosphatase (AP) > 2.5xUNL, alkaline phosphatase liver fraction must be ≤ 2.5xUNL.
  * albumin ≥ 2.5 g/dL

Exclusion Criteria:

* History of DVT or coagulation disturbances
* Need of treatment with oral anticoagulants or LMW heparin
* Clinical resistance to taxanes defined as progression during therapy or within 6 months from the end of adjuvant treatment
* Known or prior hypersensitivity to taxanes or drugs containing chemophor, or to thalidomide (or analogues)
* Preexisting peripheral neuropathy > grade 1
* Concomitant treatment with non steroid anti-inflammatory agents (NSAIA), high dose steroids or immunosuppressants
* Concomitant hormonal treatment (including those with antiandrogenic)
* Radiotherapy involving > 30% of the active bone marrow
* Radiotherapy ≤ 4 weeks prior to enrolment
* Other chemotherapy treatment ≤ 4 weeks prior to enrolment, at least 6 weeks for nitrosoureas or mitomycin C, or investigational drugs
* Symptomatic brain metastases
* Active infection
* Gastro-intestinal abnormalities, inability to take oral medication, any condition affecting absorption
* Impaired cardiac function including any of the following:

History of cardiac disease, such as myocardial infarction, in the year prior to enrollment in the clinical trial, symptomatic/uncontrolled angina pectoris, congestive heart failure or uncontrolled cardiac ischemia, or arrhythmia, abnormal left ventricular ejection fraction, or uncontrolled arterial hypertension.

* Major surgery in the two weeks prior to entering the clinical trial
* Concurrent treatment with any other anti-cancer therapy
* History of another neoplastic disease (except basal cell carcinoma of the skin or uterine cervix carcinoma in situ adequately treated), unless in remission for ≥ 5 years
* Patient unable to comply with the study protocol owing to psychological, social or geographical reasons
* Pregnant and lactating women
* Men and women of childbearing potential who are not using an effective method of contraception
* Participation in another clinical trial or treatment with any investigational product within 30 days prior to inclusion in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Define the MTD of the combination of CC-5013 and paclitaxel in patients with advanced solid tumors | 4 weeks after the first drug administration
  Number of Dose-Limiting Toxicities (DLTs)

SECONDARY OUTCOMES:
Safety profile of the drug combination | from the first administration to 30 days after the trial end
  Physical examination, laboratory and instrumental assessments and AE type and frequency
Pharmacokinetics of CC-5013 and paclitaxel given in combination | untill 4 weeks after the first drug administration
  CC-5013 and paclitaxel plasma concentration
the pharmacodynamic effects of CC-5013 and paclitaxel given in combination | from the first drug administration to 30 days after trial end
  Increase (%) in selected serum cytokines (IL2, IL6, IL10, IL12, TNFα, γIF and TGFβ).
  T-cell phenotyping:
  * T-cell markers (CD4/CD45RA/CCR7/CD3,CD8/CD45RA/CCR7/CD3)
  * Treg markers: CD4/CD25/FoxP3
  * NKcells: CD16+/CD56+
Evidence of antitumor activity in selected tumor types | From the first drug administration to 30 days after the trial end
  Response Rate according to RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Cristiana Sessa, MD, Study Chair — Istituto Oncologico della Svizzera Italiana -6500 Bellinzona, Switzerland
Locations (2):
- Fondazione IRCSS Istituto Nazionale dei Tumori, Milan, Italy
- Istituto Oncologico della Svizzera Italiana, Bellinzona, Switzerland